CLINICAL TRIAL: NCT02014883
Title: Phase II Open Label Study Using Triheptanoin in Patients With Glucose Type 1 Transporter Deficiency GLUT1-DS
Acronym: GLUT-HEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C13-37; 2013-A01300-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-12-03; First posted 2013-12-18 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2021-08

CONDITIONS: Glut1 Deficiency Syndrome
MeSH Terms: conditions — Glut1 Deficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLUT1 DS (Experimental)
  Interventions: Drug: GLUT1 DS

INTERVENTIONS:
Drug: GLUT1 DS

SUMMARY:
The purpose of this project is to study the efficacy of triheptanoin oil in patients with GLUT1 deficiency syndrome.

DETAILED DESCRIPTION:
The primary objective of the study is:

- to evaluate the capacity of triheptanoïn to improve the condition of patients with GLUT1-DS

The secondary objectives of the study are:

* to confirm the short-term safety of triheptanoïn therapy in patients with GLUT1-DS
* to evaluate the short-term effects of triheptanoïn treatment on motor function, autonomy, quality of life and clinical signs of patients with GLUT1-DS
* to evaluate the effect of triheptanoïn on brain energy metabolism using non-invasive 31P-MRS spectroscopy after activation of the occipital cortex in order to measure the levels of high-energy phosphates (such as ATP and phosphocreatine)

ELIGIBILITY:
Inclusion Criteria:

* Mutation in SLC2A1 gene
* Age > 3 years
* Patient with history/frequency of seizures or movement disorders documented at least 3 months prior to the beginning of the study
* Covered by french social security
* Patients who freely agree to participate in this study and understand the nature, risks and benefits of this study and give their written informed consent. (In addition to the requirement for the consent of parents or the legal representative, adolescents can provide additional informed consent to participate in clinical trials)

Exclusion Criteria:

* Evidence of psychiatric disorder
* Attendant neurological disorder
* Comorbid medical condition that would render them unsuitable for the study, e.g. HIV, diabetes
* Pregnant or parturient or lactating women
* Unwillingness to be informed in case of abnormal MRI
* Failure to give written informed consent
* Unable to understand the protocol
* Unable to participate to the whole study
* Absence of signed informed consent
* Persons deprived of their liberty by judicial or administrative decision
* Person subject to an exclusion period for another research
* Subjects with exclusion criteria required by french law

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Number of paroxystic events | 6 months
  The number of paroxystic events, in particular abnormal movements, will be collected during trihepatnoin treatment.

SECONDARY OUTCOMES:
Safety | 6 months
  Should the whole blood levels of propionylcarnitine increase above 8 μmol/l, the dose of triheptanoin will be reduced until the decrease of whole blood propionylcarnitine is below 8 μmol/l. Should an organic acid abnormality such as an excessive urinary excretion of propionate metabolites such as 3-hydroxypropionic, 2-methylcitric, propionylglycine, tiglylglycine and/or methylmalonic acid occur, the dose of triheptanoin will be reduced until normalization of the organic acid and acylcarnitine profile. If still abnormal, patient will be excluded from the study. For GI distress, the research dietitian will instruct the patient regarding taking the dose over a longer period of time (30 minutes). If GI distress persists, triheptanoin dose will be reduced by 50% and re-increased progressively as the problems resolve with the patients working closely with research dietitian until tolerance of the full dose is achieved.
6 minutes walk test | 6 months
9 hole Peg board | 6 months
Clinical Global Impression Scales | 6 months
Schwab-England scale | 6 months
Vineland Scale | 6 months
Fatigue Severity Scale | 6 months
Fatigue Visual Scale | 6 months
Brain 31phosphorus magnetic resonance spectroscopy | 6 months
  Ratio of Inorganic Phosphate (Pi) over Phosphocreatine during visual stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Mochel, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Brain and Spine Institute, Paris, France

REFERENCES:
- [Background] Hainque E, Meneret A, Gras D, Atencio M, Luton MP, Barbier M, De Saint Martin A, Billette de Villemeur T, Ottolenghi C, Roze E, Mochel F. Transition from ketogenic diet to triheptanoin in patients with GLUT1 deficiency syndrome. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):444-445. doi: 10.1136/jnnp-2019-321694. Epub 2019 Nov 6. No abstract available. PMID 31694879
- [Background] Hainque E, Gras D, Meneret A, Atencio M, Luton MP, Barbier M, Doulazmi M, Habarou F, Ottolenghi C, Roze E, Mochel F. Long-term follow-up in an open-label trial of triheptanoin in GLUT1 deficiency syndrome: a sustained dramatic effect. J Neurol Neurosurg Psychiatry. 2019 Nov;90(11):1291-1293. doi: 10.1136/jnnp-2018-320283. Epub 2019 Apr 4. No abstract available. PMID 30948626
- [Background] Mochel F, Hainque E, Gras D, Adanyeguh IM, Caillet S, Heron B, Roubertie A, Kaphan E, Valabregue R, Rinaldi D, Vuillaumier S, Schiffmann R, Ottolenghi C, Hogrel JY, Servais L, Roze E. Triheptanoin dramatically reduces paroxysmal motor disorder in patients with GLUT1 deficiency. J Neurol Neurosurg Psychiatry. 2016 May;87(5):550-3. doi: 10.1136/jnnp-2015-311475. Epub 2015 Nov 3. PMID 26536893